CLINICAL TRIAL: NCT05371925
Title: Endothelial Protection in Post COVID-19 Patients. The Effect of Sulodexide on Serum Levels of Biomarkers for Endothelial Dysfunction. A Prospective, Randomized, Placebo-controlled, Investigator-initiated Trial
Brief Title: Endothelial Protection in Post COVID-19 Patients With Sulodexide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Medico del Noroeste (Other)
Collaborators: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMN-01-2021
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Post COVID-19; Endothelial Dysfunction; Thrombosis
Keywords: Post COVID-19; sulodexide; thrombosis; thrombomodulin
MeSH Terms: conditions — Thrombosis | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Intervention Model Description: This is a Prospective, multicenter, randomized (1:1, placebo use) trial with a parallel-group designed
Who Masked: Participant, Care Provider, Investigator
Masking Description: participants will be randomly distributed to received either IMP or placebo at the Research site pharmacy under the same blister format and capsule appearance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulodexide group (Active Comparator): the participant will receive one Sulodexide capsule of 250LRU twice a day for 8 weeks
  Interventions: Drug: Sulodexide
- control group (Placebo Comparator): the participant will receive on placebo capsule twice a day for 8 weeks of same appearance as IMP
  Interventions: Drug: Sulodexide

INTERVENTIONS:
Drug: Sulodexide — one 250LRU sulodexide capsule twice a day for 8 weeks
  Other Names: Vessel due F (Alfasgima SpA, Italy)

SUMMARY:
This is a Prospective, multicenter, randomized (1:1, placebo use) trial with a parallel-group design to assess if the use of sulodexide influences serum levels of biomarkers for endothelial dysfunction on convalescent COVID-19 patients who suffered a moderate (or more severe) clinical presentation and have chronic comorbidities of high risk for endothelial dysfunction.

The recruitment period is estimated at 6 months. The follow-up period of all participants will be 8 weeks.

The participant will receive according to group allocation after randomization

1. study group: sulodexide oral dose of 250LRU capsule bid for 8 weeks.
2. control group: placebo oral dose of 1 capsule bid for 8 weeks.

Participants in both groups will continue the standard of care recommended by national healthcare guidelines for each Country, including any concomitant medication indicated by their primary physician.

DETAILED DESCRIPTION:
Background Endothelial cells play an important role in SARS-CoV-2 infection, not only as target organs but also as effectors, with several pathways possibly involved, all more widely analyzed in the acute phase. However, the exact mechanism of post-COVID-19 cardiovascular events is not fully understood nor is its involvement in perpetuating a chronic proinflammatory and prothrombotic state. Sulodexide has many useful pleitropic properties where the restoration of a proper functional endothelium should be a paramount objective to achieve when possible.

Design This is a Prospective, multicenter, randomized (1:1, placebo use) trial with a parallel-group design to assess if the use of sulodexide influences serum levels of biomarkers for endothelial dysfunction on convalescent COVID-19 patients who suffered a moderate (or more severe) clinical presentation and have chronic comorbidities of high risk for endothelial dysfunction.

The recruitment period is estimated at 6 months. The follow-up period of all participants will be 8 weeks.

The participant will receive according to group allocation after randomization

1. study group: sulodexide oral dose of 250LRU capsule bid for 8 weeks.
2. control group: placebo oral dose of 1 capsule bid for 8 weeks. Participants in both groups will continue the standard of care recommended by national healthcare guidelines for each Country, including any concomitant medication indicated by their primary physician.

Participation in the trial is strictly voluntary. Patients, relatives, or the scientific guardian can withdraw his/her consent at any time without giving further explanation, and without prejudice to further medical care and treatment.

All concomitant therapies will be permitted for the patients to receive full supportive care during the study, as appropriate. For the purpose of the study, relevant concomitant treatment received during the study, including those for COVID-19, will be recorded in the CRF.

Other anticoagulant drugs are not permitted within 1 day of screening. If criteria for participation are met, the patient will wait 5 days to start the protocol process.

If the patients during the course of the trial are in need of prophylactic low-dose anticoagulation, patients will be closely monitored for any bleeding complications. If full-dose anticoagulation is needed, sulodexide will be suspended, but the patients will not be excluded.

The Sponsor is responsible for setting up the randomization system. The randomization sequence will be done in permuted blocks of variable sizes stratified for a trial site using centralized, concealed allocation.

The following assessments will be performed at each participating research center to determine eligibility requirements, as specified in the selection criteria:

* recorded laboratory-confirmed SARS-CoV-2 infection as determined by PCR in naso/oropharyngeal swabs or any other relevant specimen obtained during the course of the disease. Alternative tests (e.g., rapid antigenic tests) are also acceptable as laboratory confirmation is their specificity has been accepted by the Sponsor.
* Focused medical history, including the following information: Date of onset of COVID-19 symptoms (fever and/or other symptoms). History of chronic medical conditions related to the selection criteria or known risk factors for COVID-19. Confirm hospitalization/ICU admission period/duration due to COVID.

The overall eligibility of the subject to participate in the study will be assessed once all screening data are available. The screening process can be suspended prior to completing the assessment at any time if exclusions are identified by the research team. Study subjects who qualify will be immediately randomized after the informed consent is signed, and scheduled for a blood sample test at the earliest convenience. Oral medication will start after the blood sample has been taken.

If allocated to the study group, the patient will receive an oral dose of 250LRU twice daily for 8 weeks. If allocated to the control group, the patient will receive an oral dose of placebo in a similar appearance to sulodexide twice daily for 8 weeks.

Screening (Day - 3/ -1) participants will be screened for selection criteria. A signed informed consent form will be obtained, clinical history, Health risk calculator, concomitant medication, and inclusion/exclusion criteria will be assessed. If eligible to participate the subject will proceed to the randomization process and be scheduled for a blood sample test at the earliest convenience. The participant will continue the standard of care established by their primary physician

Visit 1 (Day 1) patients will present to the research site, verification of complete information gathered at screening (clinical history, concomitant medication, inclusion/exclusion criteria, and signed informed consent) if missing data is detected this will be completed. The patient will receive a physical examination including vital signs and be escorted to have a blood sample taken at the research site laboratory. A baseline evaluation of thrombotic/thromboembolic events, the WHO ordinal clinical progression scale, and the Post Covid-19 functional status will be performed. Any adverse event will also be evaluated.

After blood sample results is taken, the patient will start the oral dose of the study medication or placebo according to group allocation. The participant will be free to contact the research site for any doubts or comments regarding the trial and schedule an extra visit if deemed necessary. The patient will continue the standard of care for the COVID-19 convalescent process under the management of the participant healthcare provider.

Follow-up visit 1 (week 4) where adverse events will be evaluated, as of medication compliance. Physical examination including vital signs will be performed, and concomitant medication recorded. The presence of any relevant clinical symptoms will be addressed. A blood sample test will be taken (laboratory assessments are described in section 11.2). Thrombotic/thromboembolic events, the WHO 10-point ordinal clinical progression scale, and the Post-COVID functional status will be assessed.

Follow-up visit 2 (week 8) where adverse events will be evaluated, as of medication compliance. Physical examination including vital signs will be performed, and concomitant medication recorded. The presence of any relevant clinical symptoms will be addressed. A blood sample test will be taken (laboratory assessments are described in section 11.2). Thrombotic/thromboembolic events, the WHO 10-point ordinal clinical progression scale, and the post-COVID functional status will be assessed. At this time, the patient participation in the trial will end.

Data Analysis

The definitions of trial populations are as follows:

Intention-to-treat This will comprise all randomized patients (except those randomized in error who never received the trial medication). This population will be evaluated for all endpoints Per -protocol This is a subset of the intention-to-treat population encompassing correctly included patients who have received sulodexide or Placebo according to the protocol. This population will be evaluated for the primary endpoint only.

Continuous variables will be expressed as mean and standard deviation and compared using the Student's T-test; categorical variables will be compared with the Chi-square test or the Fisher exact test. Values of p less than 0.05 will be considered statistically significant.

Proportions will be compared between the two intervention-arms within each group using the Fisher exact test and presented as relative risk ratio (RR) or reduction of the RR (1- RR *100%) if RR lower than 1. Adjustment for covariates and possible confounders will be done using Poisson regression with a log link and robust estimate of the covariance (Huber method), using the method proposed by Zou et al. 2014 and 2013. Continuous variables will be compared between groups using Wilcoxon rank-sum test and the effect presented as Mean Difference. Adjustment for covariates and possible cofounders will be done using ordinary least square regression. Variables will be transformed to the logarithm scale if normality is improved, and results presented as Proportional Difference. If after transformation, the non-normality of the residuals is detected using diagnostic regression plots, robust intervals of confidence and Wald test will be presented instead.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* male or female
* Patients with documented PCR SARS-CoV-2 positive test obtained during the course of the disease
* Convalescent COVID-19 patient (define as at least 10 days after the onset of symptoms, no fever for at least 24 hours without the use of antipyretics and improvement of respiratory symptoms according to the quick COVID-19 Severity Index (qCSI).
* Signature of informed consent.
* moderate or worst clinical severity presentations of COVID-19. (According to the World Health Organization Clinical progression scale)
* Risk of health complication >50% according to the Health risk calculator

Exclusion Criteria:

* concomitant use of another anticoagulant.
* known pregnancy.
* known hypersensitivity to sulodexide
* the need for hospital care at screening
* Renal insufficiency with CrCl <30ml/min or continuous renal replacement therapy, hemodialysis, or peritoneal dialysis.
* Blood platelet count < 30 000/µL
* Other conditions that are judged to carry an increased risk of bleeding as judged by the investigator

Elimination criteria:

A patient randomized in error (monitoring shows that in- or exclusion criteria have been violated) who never received the trial medication, will be excluded from all analyses

The investigator must discontinue study treatment for a given patient at any time for the following reasons:

• In case of intolerable serious adverse reactions/events, which are clinically relevant, suspected to be related to trial intervention, and affect the patient´s safety. This will be at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
thrombomodulin | compare baseline level at 4 weeks of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum thrombomodulin levels compared to placebo use.
thrombomodulin | compare baseline level at 8 weeks of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum thrombomodulin levels compared to placebo use.

SECONDARY OUTCOMES:
P-Selectin | compare baseline level to the ones at 4 weeks of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum P-Selectin levels compared to placebo use.
P-Selectin | compare baseline level to the ones at 8 weeks of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum P-Selectin levels compared to placebo use.
Troponin I | compare baseline level to the ones at 4 weeks of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum Tissue factor levels compared to placebo use.
Troponin I | compare baseline level to the ones at 8 weeks of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum Tissue factor levels compared to placebo use.
Von Willebrand factor | compare baseline level to the ones at 4 weeks of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum Von Willebrand factor levels compared to placebo use.
Von Willebrand factor | compare baseline level to the ones at 8 weeks of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum Von Willebrand factor levels compared to placebo use.
ICAM-1 | compare baseline level to the ones at 4 week and 8 week of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum ICAM-1 levels compared to placebo use.
VCAM-1 | compare baseline level to the ones at 4 week and 8 week of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum VCAM-1 levels compared to placebo use.
D-dimer | compare baseline level to the ones at 4 week and 8 week of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum D-dimer levels compared to placebo use.
C reactive protein | compare baseline level to the ones at 4 week and 8 week of treatment
  Assess whether the use of sulodexide in convalescent COVID-19 patients affects serum C-reactive protein levels compared to placebo use.

OTHER OUTCOMES:
post-COVID-19 functional status | compare at 4 week and 8 week of treatment
  Evaluate whether there is a difference in clinical progression of the disease in convalescent COVID-19 patients, according to the post-COVID-19 functional status scale grade with the use of sulodexide compared to placebo.
the WHO clinical progression | compare at 4 week and 8 week of treatment
  Evaluate whether there is a difference in clinical progression of the disease in convalescent COVID-19 patients, according to the WHO clinical progression scale with the use of sulodexide compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro J Gonzalez-Ochoa, MD, Principal Investigator — Centro Medico del Noroeste
Locations (1):
- Centro Medico del Noroeste, San Luis Río Colorado, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No